CLINICAL TRIAL: NCT03860974
Title: A Randomized, Subject-Masked, Active-Controlled, Parallel-Arm Clinical Trial Comparing Serratus Plane and Paravertebral Nerve Blocks
Brief Title: Serratus Plane Versus Paravertebral Nerve Blocks for Breast Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Brian M. Ilfeld, MD, MS, Professor of Anesthesiology, In Residence, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Serratus vs PVB
Record Dates: First submitted 2019-02-28; First posted 2019-03-04 (Actual); Results first posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-08

CONDITIONS: Breast Surgery
Keywords: regional anesthesia; paravertebral; erector spinae; nerve block
MeSH Terms: interventions — Injections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Serratus Plane (single injection) (Experimental): A single injection serratus plane block will be administered using ropivacaine 0.5% with epinephrine 1:200,000-400,000 (20 mL for unilateral surgery; 16 mL on each side for bilateral surgery)
  Interventions: Drug: Serratus Plane block (single injection)
- Paravertebral (single injection) (Active Comparator): Single injection paravertebral blocks will be administered using ropivacaine 0.5% with epinephrine 1:200,000-400,000 (20 mL for unilateral surgery; 16 mL each side for bilateral surgery)
  Interventions: Drug: Paravertebral block (single injection)

INTERVENTIONS:
Drug: Serratus Plane block (single injection) — A single-injection serratus plane block will be administered using ropivacaine 0.5% with epinephrine 1:200,000-400,000 (20 mL of local anesthetic for unilateral surgery; 16 mL of local anesthetic each side for bilateral surgery).
  Arms: Serratus Plane (single injection)
Drug: Paravertebral block (single injection) — Single injection paravertebral blocks will be administered using ropivacaine 0.5% with epinephrine 1:200,000-400,000 (20 mL for unilateral surgery; 16 mL each side for bilateral surgery). For paravertebral blocks without axillary involvement, this will be at the T3 and T5 levels. For paravertebral blocks with axillary involvement, this will be at the T2 and T4 levels. For unilateral PVBs, 10 mL of local anesthetic will be injected per level. For bilateral paravertebral blocks, 8 mL of local anesthetic will be injected per level.
  Arms: Paravertebral (single injection)

SUMMARY:
Following painful surgical procedures of the breast, postoperative analgesia is often provided with a paravertebral nerve block (PVB). For intense, but shorter-duration acute pain, a single-injection of local anesthetic is used with a duration of approximately 12 hours. Recently an alternative block has been reported: the serratus plane block.2 The theoretical benefits include ease of administration since it is a plane superficial to the PVB and therefore easier to identify and target with ultrasound (therefore increasing success rate); and an increased safety margin as there are fewer anatomic structures in the immediate area which could be injured with the needle; and, the target plane is much further from the intrathecal/epidural space relative to the PVB, therefore leakage of cerebrospinal fluid or injury to the spinal cord are less likely with the serratus compared to the PVB.3 There are, therefore, multiple theoretical reasons to prefer the serratus over the PVB. Unfortunately, it remains unknown if the analgesia provided by this new technique is comparable to that provided with the PVB.4 The investigators therefore propose to compare these two techniques with a randomized, subject-masked, active-controlled, parallel-arm clinical trial.

DETAILED DESCRIPTION:
This investigation will be a randomized, subject-masked, active-controlled parallel-arm, human subjects clinical trial. Of note, the investigators will be using standard-of-care local anesthetic under an FDA-approved purpose and do not plan to research a possible change of indication or use of these medications as part of this research project. The treatments in both groups are currently used at our institution and there is true clinical equipoise at this time. The only difference in treatment between subjects who enroll versus those not enrolled in this study will be those who enroll will have the decision between which anatomic block location determined randomly, as opposed to the physician simply choosing him/herself.

Enrollment. Consenting adults undergoing breast surgery with a planned single-injection regional analgesic will be offered enrollment. Patients undergoing breast surgery with a planned perineural catheter regional analgesic will be excluded. Study inclusion will be proposed to eligible patients prior to surgery. If a patient desires study participation, written, informed consent will be obtained using a current UCSD IRB-approved ICF. Selection for inclusion will not be based on gender, race, or socioeconomic status. The study population of interest includes men and women of all races and socioeconomic status.

Preoperative Procedures. Following written, informed consent, the investigators will collect baseline anthropomorphic information (e.g., age, sex, height, and weight). All subjects will have a peripheral intravenous (IV) catheter inserted, standard noninvasive monitors applied, supplemental oxygen administered via a nasal cannula or face mask, and placed in the sitting position. Midazolam and fentanyl (IV) will be titrated for patient comfort, while ensuring that patients remain responsive to verbal cues. Both possible block locations will be viewed with ultrasound. If one or both of the locations is unacceptable for block placement in the clinician's opinion, the subject will not be randomized and will not proceed further with the study.

Subjects will then be randomized using a computer-generated list and opaque, sealed envelopes to one of two treatment groups: (blocks of 4, stratified for unilateral vs. bilateral surgery): (1) serratus plane or (2) paravertebral block. All blocks will be placed by a regional anesthesia fellow or resident under the direct supervision and guidance of a regional anesthesia attending (or by the attending themselves).

The area of needle insertion will be cleaned with chlorhexidine gluconate and isopropyl alcohol. All blocks will be placed using standard UCSD ultrasound-guided techniques as previously described.

Ropivacaine 0.5% (20 mL for unilateral surgery; 16 mL each side for bilateral surgery) will be administered via the needle into the target plane(s). For PVBs without axillary involvement, this will be at the T3 and T5 levels. For PVBs with axillary involvement, this will be at the T2 and T4 levels. For unilateral PVBs, 10 mL of local anesthetic will be injected per level. For bilateral PVBs, 8 mL of local anesthetic will be injected per level.

Single-injection blocks will be considered successful if, within 30 minutes, the subject experiences decreased sensation to cold temperature with an alcohol pad over the approximate level of the ipsilateral 4th thoracic dermatome. Misplaced blocks will be replaced successfully, or the patient excluded from further study participation. For subjects undergoing bilateral surgical procedures, a block using the same protocol will be administered on the contralateral side.

Intraoperatively, all subjects will receive a general anesthetic using inhaled and intravenous anesthetic and oxygen. Intravenous fentanyl will be administered for cardiovascular responsiveness to noxious stimuli at the discretion of the anesthesia provider.

Postop: Subjects will be discharged with a prescription for oxycodone 5 mg tablets for supplementary analgesia and instructed to record the time at which they take their first opioid tablet as well as the time at which they believe the block starts to wear off.

Outcome measurements (end points). Pain scores will be recorded using the NRS. Within the recovery room, pain scores, opioid requirements, and antiemetic administration will be recorded by nursing staff masked to treatment group. The morning following surgery, all subjects will be contacted by phone or in person [if hospitalized] to record lowest, average, highest, and current pain scores; sleep disturbances, and nausea using a 0-10 Likert scale (0 = no nausea; 10 = vomiting). For outpatients, opioid requirements will be recorded while inpatients will have opioid requirements extracted from the electronic medical record. In addition, the investigators will extract antiemetic use from the electronic record. They will collect the times at which subjects felt their block resolve and they consumed their first opioid analgesic pills following recovery room discharge.

Hypothesis 1: Following breast surgery, analgesia will be non-inferior in the recovery room with a serratus plane block compared with a paravertebral block as measured with the Numeric Rating Scale.

Hypothesis 2: For breast surgery, opioid consumption will be non-inferior in the operating and recovery rooms with a serratus plane block compared with a paravertebral block (primary: cumulative intravenous morphine equivalents).

Primary end point: In order to claim that serratus plane blocks are non-inferior to paravertebral blocks, both Hypotheses 1 and 2 must be at least non-inferior.

Statistical methods. Descriptive statistics will be provided by arm and in aggregate. Baseline characteristics of arms will be compared using the Wilcoxon-Mann-Whitney and Fisher's Exact tests. Key characteristics that are significantly different (p<0.05) will be included as covariates in the analysis models.

Primary aim. The investigators will test the noninferiority of the serratus nerve block compared to the paravertebral nerve block. The 95% confidence interval (CI) associated with the Wilcoxon-Mann-Whitney test will be derived for the group difference (paravertebral minus serratus) in median pain scores within the recovery room. If the lower limit of the 95% CI is greater than -1.25, the investigators will conclude noninferiority. If there are significant differences between the groups in any key characteristics, these characteristics will be included as covariates in a linear model. The same noninferiority margin (-1.25) will be applied to the 95% CI for the covariate adjusted group difference in mean pain derived from the linear model.

The noninferiority of the serratus nerve block with regard to total opioid consumption within the operating and recovery rooms will be tested in the same manner as pain, i.e. comparing the limits of a 95% CI associated with the Wilcoxon-Mann-Whitney test to a predefined noninferiority margin (in this case 2 mg). Covariate adjusted linear models will again be applied in the event that key characteristics are significantly different between the groups.

Sample size justification. Power for the Wilcoxon-Mann-Whitney derived noninferiority testing is based on 10,000 simulated trials. The investigators simulated pain scores from a discrete distribution with median (interquartile range) 3 (2-5). Between the quartiles, the probability of each score was assumed constant. The distribution for each group was assumed to be the same. The sample size of n=50 per group provides 82% power to detect noninferiority in pain with a margin of 1.25. Similarly, opioid consumption was assumed to follow a truncated normal distribution with mean 2.5 mg and standard deviation 2 mg, and minimum value 0 mg. The sample size of n = 50 per group provides at least 95% power to detect noninferiority with margin 2 mg. Therefore, the investigators will enroll 50 subjects for each of two treatments with primary end point values for a total enrollment of 100 subjects with a primary end point. To allow for dropouts, the investigators will request a maximum enrollment of 120 subjects. Noninferiority in pain is tested first, and if significant, noninferiority in opioid consumption is tested. Under this hierarchical testing framework, no adjustment in alpha is necessary to control Type 1 error.

ELIGIBILITY:
Inclusion Criteria:

* undergoing unilateral or bilateral breast surgery with at least moderate postoperative pain anticipated
* analgesic plan includes a single-injection peripheral nerve block(s)
* age 18 years or older

Exclusion Criteria:

* morbid obesity as defined by a body mass index > 40 (BMI=weight in kg / [height in meters]2)
* renal insufficiency (preoperative creatinine > 1.5 mg/dL)
* chronic opioid use (daily use within the 2 weeks prior to surgery and duration of use > 4 weeks)
* history of opioid abuse
* any comorbidity which results in moderate or severe functional limitation inability to communicate with the investigators or hospital staff
* pregnancy
* planned regional analgesic with perineural catheter placement
* incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2021-02-12 (Actual); Study Completion 2021-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Ilfeld, MD, MS, Principal Investigator — UCSD Medical Center
Locations (1):
- University California San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gabriel RA, Swisher MW, Sztain JF, Curran BP, Said ET, Abramson WB, Khatibi B, Alexander BS, Finneran JJ, Wallace AM, Armani A, Blair S, Dobke M, Suliman A, Reid C, Donohue MC, Ilfeld BM. Serratus anterior plane versus paravertebral nerve blocks for postoperative analgesia after non-mastectomy breast surgery: a randomized controlled non-inferiority trial. Reg Anesth Pain Med. 2021 Sep;46(9):773-778. doi: 10.1136/rapm-2021-102785. Epub 2021 Jun 22. PMID 34158376

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Serratus Plane (Single Injection) | Paravertebral (Single Injection)
Started | 49 | 51
Completed | 49 | 51
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Serratus: Ropivacaine 0.5% (20 mL for unilateral surgery; 16 mL each side for bilateral surgery) will be administered via the needle into the target plane(s). For serratus blocks, local anesthetic will be deposited above rib 5 and deep to serratus muscle in the lateral position.
- Paravertebral: Ropivacaine 0.5% (20 mL for unilateral surgery; 16 mL each side for bilateral surgery) will be administered via the needle into the target plane(s). For PVBs without axillary involvement, this will be at the T3 and T5 levels. For PVBs with axillary involvement, this will be at the T2 and T4 levels. For unilateral PVBs, 10 mL of local anesthetic will be injected per level. For bilateral PVBs, 8 mL of local anesthetic will be injected per level.
- Total: Total of all reporting groups
Arm/Group | Serratus | Paravertebral | Total
Number analyzed (Participants) | 49 | 51 | 100
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 55 [44 to 64] | 53 [41.5 to 61.5] | 53 [41.5 to 61.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 48 | 97
  Male | 0 | 3 | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 49 | 51 | 100

OUTCOME MEASURES:

1. Primary Outcome: Mean/Median Numeric Rating Scale Pain Score Within the Recovery Room
Description: Numeric Rating Scale: the NRS is a segmented numeric version of the Visual Analog Scale (VAS) in which the study subject selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. This 11-point numeric scale ranges from 0 representing "no pain" to 10 representing "worst imaginable pain." Higher numeric scores represent increased pain and thus worse outcomes. The primary outcome measure will be the mean or median (depending on whether data is normally or not normally distributed) of all reported NRS within the recovery room following surgery and prior to recovery room discharge.
Time Frame: Within the recovery room, averaging approximately 2 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Serratus Plane (Single Injection) | Paravertebral (Single Injection)
Number analyzed (Participants) | 49 | 51
score on a scale | 4 [0 to 5.5] | 0 [0 to 3.0]
Statistical Analysis 1: Comparison: Serratus Plane (Single Injection) vs Paravertebral (Single Injection); Test type: Non-Inferiority — We tested the non-inferiority of serratus block compared with PVB using the 95% CI associated with the Wilcoxon-Mann-Whitney test with continuity correction. If the lower limit of the 95% CI for median "average" PACU pain scores was greater than -1.25 , we would conclude non-inferiority. The non-inferiority of serratus blocks with regard to opioid consumption was similarly tested to a predefined non-inferiority margin of 2 mg intravenous morphine equivalents; p = 0.001, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 4

2. Secondary Outcome: Number of Participants Requiring an Anti-emetic Within the Recovery Room
Description: This outcome is measured based on whether the patient needed an anti-emetic in the recovery room following surgery and prior to discharge from the recovery room. An "anti-emetic" is a medication given if the patient complains of nausea or exhibits vomiting.
Time Frame: Within the recovery room, averaging approximately 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Serratus Plane (Single Injection) | Paravertebral (Single Injection)
Number analyzed (Participants) | 49 | 51
Participants | 19 | 8

3. Secondary Outcome: Opioid Consumption After Recovery Room Discharge
Description: cumulative opioid consumed between the recovery room discharge to the postoperative day 1 data collection phone call measured in morphine milliequivalents
Time Frame: Between the recovery room discharge to the postoperative day 1 data collection phone call
Measure: Median (Inter-Quartile Range); unit: mg in morphine equivalents
Arm/Group | Serratus Plane (Single Injection) | Paravertebral (Single Injection)
Number analyzed (Participants) | 49 | 51
mg in morphine equivalents | 2 [2 to 4] | 2 [0 to 4]

4. Secondary Outcome: WORST Pain Measured Using the Numeric Rating Scale Pain Score
Description: Numeric Rating Scale: the NRS is a segmented numeric version of the Visual Analog Scale (VAS) in which the study subject selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. This 11-point numeric scale ranges from 0 representing "no pain" to 10 representing "worst imaginable pain." Higher numeric scores represent increased pain and thus worse outcomes. This outcome was the "worst" pain experienced by the patient Between the recovery room discharge to the postoperative day 1 data collection phone call as reported during that data collection phone call.
Time Frame: Between the recovery room discharge to the postoperative day 1 data collection phone call
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Serratus Plane (Single Injection) | Paravertebral (Single Injection)
Number analyzed (Participants) | 49 | 51
score on a scale | 5 [3 to 6] | 3 [2 to 5]

5. Secondary Outcome: Lowest Pain Measured Using the Numeric Rating Scale Pain Score
Description: Numeric Rating Scale: the NRS is a segmented numeric version of the Visual Analog Scale (VAS) in which the study subject selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. This 11-point numeric scale ranges from 0 representing "no pain" to 10 representing "worst imaginable pain." Higher numeric scores represent increased pain and thus worse outcomes. This outcome was the "least" pain experienced by the patient between the recovery room discharge to the postoperative day 1 data collection phone call as reported during that data collection phone call.
Time Frame: between the recovery room discharge to the postoperative day 1 data collection phone call
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Serratus Plane (Single Injection) | Paravertebral (Single Injection)
Number analyzed (Participants) | 49 | 51
units on a scale | 1 [0 to 3] | 0 [0 to 1]

6. Secondary Outcome: Average Pain Measured Using the Numeric Rating Scale Pain Score
Description: Numeric Rating Scale: the NRS is a segmented numeric version of the Visual Analog Scale (VAS) in which the study subject selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. This 11-point numeric scale ranges from 0 representing "no pain" to 10 representing "worst imaginable pain." Higher numeric scores represent increased pain and thus worse outcomes. This outcome was the "average" pain experienced by the patient between the recovery room discharge to the postoperative day 1 data collection phone call as reported during that data collection phone call.
Time Frame: between the recovery room discharge to the postoperative day 1 data collection phone call
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Serratus Plane (Single Injection) | Paravertebral (Single Injection)
Number analyzed (Participants) | 49 | 51
score on a scale | 3 [2 to 4] | 2 [0.5 to 3]

7. Secondary Outcome: Worst RECOVERY ROOM Pain Measured Using the Numeric Rating Scale Pain Score
Description: Numeric Rating Scale: the NRS is a segmented numeric version of the Visual Analog Scale (VAS) in which the study subject selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. This 11-point numeric scale ranges from 0 representing "no pain" to 10 representing "worst imaginable pain." Higher numeric scores represent increased pain and thus worse outcomes. This outcome was the highest/maximum pain score reported by the patient within the recovery room.
Time Frame: within the recovery room following surgery and prior to recovery room discharge
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Serratus Plane (Single Injection) | Paravertebral (Single Injection)
Number analyzed (Participants) | 49 | 51
units on a scale | 5 [3 to 6] | 3 [2 to 5]

8. Secondary Outcome: Awakenings Due to Pain
Description: The number of times the subject recalls awakening from sleep due to pain the prior evening
Time Frame: the first evening after surgery, averaging approximately 8 hours
Measure: Median (Inter-Quartile Range); unit: number of awakenings
Arm/Group | Serratus Plane (Single Injection) | Paravertebral (Single Injection)
Number analyzed (Participants) | 49 | 51
number of awakenings | 0 [0 to 0] | 0 [0 to 0]

9. Primary Outcome: Mean/Median Opioid Consumption Within the Recovery Room
Description: Opioid consumption as measured in milligram morphine equivalents. The primary outcome measure will be the mean or median (depending on whether data is normally or not normally distributed) of the cumulative opioid consumption within the recovery room following surgery and prior to recovery room discharge.
Time Frame: Within the recovery room following surgery and prior to recovery room discharge
Measure: Median (Inter-Quartile Range); unit: milligrams of morphine equivalents
Arm/Group | Serratus Plane (Single Injection) | Paravertebral (Single Injection)
Number analyzed (Participants) | 49 | 51
milligrams of morphine equivalents | 14 [10 to 19] | 10 [10 to 16]

10. Secondary Outcome: LEAST RECOVERY ROOM Pain Measured Using the Numeric Rating Scale Pain Score
Description: Numeric Rating Scale: the NRS is a segmented numeric version of the Visual Analog Scale (VAS) in which the study subject selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. This 11-point numeric scale ranges from 0 representing "no pain" to 10 representing "worst imaginable pain." Higher numeric scores represent increased pain and thus worse outcomes. This outcome was the lowest pain score reported by the patient within the recovery room.
Time Frame: within the recovery room following surgery and prior to recovery room discharge
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Serratus Plane (Single Injection) | Paravertebral (Single Injection)
Number analyzed (Participants) | 49 | 51
units on a scale | 0 [0 to 3] | 0 [0 to 1]

11. Secondary Outcome: Opioid Consumption Within the Operating Room
Description: cumulative opioid consumed between entry into the operating room and discharge to the recovery room as measured in morphine milliequivalent
Time Frame: Within the operating room, averaging approximately 2 hours
Measure: Median (Inter-Quartile Range); unit: mg in morphine equivalents
Arm/Group | Serratus Plane (Single Injection) | Paravertebral (Single Injection)
Number analyzed (Participants) | 49 | 51
mg in morphine equivalents | 10 [10 to 10] | 10 [8.75 to 10]

12. Secondary Outcome: Nausea and Vomiting Following Recovery Room Discharge
Description: A likert scale was used in which 0 represented no nausea experienced, and 10 represented active vomiting.
Time Frame: between discharge from the recovery room and the data collection phone call on postoperative day 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Serratus Plane (Single Injection) | Paravertebral (Single Injection)
Number analyzed (Participants) | 49 | 51
units on a scale | 0 [0 to 0] | 0 [0 to 0]

13. Secondary Outcome: Time From Recovery Room Discharge Until First Opioid Use
Description: The time in hours between recovery room discharge and the first use of an opioid as reported by patients during the data collection phone call on postoperative day 1. For patients who did not consume any opioids following recovery room discharge, their time was recorded as 24 hours for calculation purposes.
Time Frame: between discharge from the recovery room and the data collection phone call on postoperative day 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Serratus Plane (Single Injection) | Paravertebral (Single Injection)
Number analyzed (Participants) | 49 | 51
hours | 14 (4) | 8 (1)

14. Secondary Outcome: Time From Recovery Room Discharge Until Block Resolution
Description: The time in hours between local anesthetic injection completion during the nerve block and the time when block resolution began as reported by patients during the data collection phone call on postoperative day 1.
Time Frame: between local anesthetic injection completion during the nerve block and the time when block resolution began
Population: ** This outcome was erroneously left off of the case report forms, so we did not collect the data for this outcome measure.
Arm/Group | Serratus Plane (Single Injection) | Paravertebral (Single Injection)
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: WORST Pain Measured DURING NERVE BLOCK Using the Numeric Rating Scale Pain Score
Description: Numeric Rating Scale: the NRS is a segmented numeric version of the Visual Analog Scale (VAS) in which the study subject selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. This 11-point numeric scale ranges from 0 representing "no pain" to 10 representing "worst imaginable pain." Higher numeric scores represent increased pain and thus worse outcomes. This outcome was the "worst" pain experienced by the patient during the placement of the nerve block between the time the block needle was inserted until the time the block needle was withdrawn.
Time Frame: During the placement of the nerve block
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Serratus Plane (Single Injection) | Paravertebral (Single Injection)
Number analyzed (Participants) | 49 | 51
score on a scale | 2 [0 to 4] | 1 [1 to 3.5]

16. Secondary Outcome: Average Pain Measured DURING NERVE BLOCK Using the Numeric Rating Scale Pain Score
Description: Numeric Rating Scale: the NRS is a segmented numeric version of the Visual Analog Scale (VAS) in which the study subject selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. This 11-point numeric scale ranges from 0 representing "no pain" to 10 representing "worst imaginable pain." Higher numeric scores represent increased pain and thus worse outcomes. This outcome was the "average" pain experienced by the patient during the placement of the nerve block between the time the block needle was inserted until the time the block needle was withdrawn.
Time Frame: During the placement of the nerve block
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Serratus Plane (Single Injection) | Paravertebral (Single Injection)
Number analyzed (Participants) | 49 | 51
score on a scale | 1 [0 to 2] | 1 [0 to 2]

17. Secondary Outcome: Time to Perform Nerve Block
Description: The time in minutes between the time from initial nerve block needle insertion until nerve block needle withdrawal, measured in minutes.
Time Frame: The time from initial nerve block needle insertion until nerve block needle withdrawal
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Serratus Plane (Single Injection) | Paravertebral (Single Injection)
Number analyzed (Participants) | 49 | 51
minutes | 1.25 [0 to 4] | 4 [2 to 6]

ADVERSE EVENTS:
Time Frame: up to 24 hours after surgery
Arm/Group | Serratus Plane (Single Injection) | Paravertebral (Single Injection)
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/51
Other Adverse Events (participants affected / at risk) | 0/49 | 0/51

LIMITATIONS AND CAVEATS:
** Regarding the time from nerve block placement until block resolution, this outcome was erroneously left off of the case report forms, so we did not collect the data for this outcome measure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-01): https://cdn.clinicaltrials.gov/large-docs/74/NCT03860974/Prot_SAP_002.pdf